CLINICAL TRIAL: NCT05335642
Title: Secondary Intervention and Surveillance After Abdominal Aortic Aneurysm Endovascular Repair: Retrospective Cohort Study
Brief Title: Secondary Intervention and Surveillance After EVAR
Status: Completed | Type: Observational
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Marina Felicidade Dias Neto, Principal Investigator, Hospital Sao Joao
Other Study IDs: 10353
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Patients that had secondary interventions after EVAR
  Interventions: Procedure: EVAR
- Patients without secondary interventions after EVAR
  Interventions: Procedure: EVAR

INTERVENTIONS:
Procedure: EVAR — Endovascular repair of abdominal aortic aneurysms

SUMMARY:
This is a retrospective cohort study of consecutive patients submitted to elective EVAR, between February/2009 and May/2019 in a single institution. Symptomatic or ruptured AAA, mycotic aneurysms, isolated iliac aneurysms and complex abdominal aortic repairs were excluded. The primary outcomes were freedom from secondary intervention and compliance with follow-up, defined as surveillance imaging performed within a periodicity no longer than 18 months.

ELIGIBILITY:
Inclusion Criteria:

* This is a retrospective cohort study of consecutive patients submitted to elective EVAR, between February/2009 and May/2019 in a single institution.

Exclusion Criteria:

* Symptomatic or ruptured AAA, mycotic aneurysms, isolated iliac aneurysms and complex abdominal aortic repairs were excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients submitted to elective EVAR in a university center.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participant with secondary intervention (SI) after EVAR | 5 years follow up
  SI included: access-related SI included suture of access bleeds, distal thrombo-embolectomy, patch angioplasty, or thromboendarterectomy of the common femoral artery; limb graft occlusion was defined as a thrombotic obstruction of blood flow in one or both endograft limbs, being a potential threat to the limb; lower limb ischemia was considered when there was a decrease in arterial perfusion of the limb, that was not related with limb graft occlusion; endoleak; stent migration was reported if no simultaneous type 1 endoleak was observed.

SECONDARY OUTCOMES:
Number of participant with compliance with follow-up after EVAR | 5 years follow up
  Non-compliance with surveillance was defined by an 18 months period in which no surveillance imaging was performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Marina Felicidade Dias Neto, Porto, State/Province, Portugal

IPD SHARING:
Plan to Share IPD: Undecided